CLINICAL TRIAL: NCT01745731
Title: Clinical Trial Phase II Multicenter Open Randomized Trial of the Therapeutic Use of Cells Intraportal Infusion of Autologous Bone Marrow Mononuclear as Enhancing Liver Regeneration Prior to Performing Extended Hepatic Resection.
Brief Title: Cell Infusion Intraportal Autologous Bone Marrow Mononuclear as Enhancer of Liver Regeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Iniciativa Andaluza en Terapias Avanzadas (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMMo/RH/2009; 2009-017793-20 (EudraCT Number)
Record Dates: First submitted 2012-12-03; First posted 2012-12-10 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Liver Transplant Rejection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Patients with hepatic space occupying lesion requiring an extended hepatic resection to those who were preoperatively performed a Cell infusion intraportal mononuclear bone marrow autologous and portal embolization of the affected segments.
  Interventions: Other: Cell infusion intraportal mononuclear bone marrow autologous and portal embolization of the affected segments.
- Control (No Intervention): Patients with hepatic space occupying lesion that require an extended liver resection that were performed preoperatively portal embolization of the affected segments.

INTERVENTIONS:
Other: Cell infusion intraportal mononuclear bone marrow autologous and portal embolization of the affected segments. — Proceeds to selective application of stem cells in the portal branches of segments II and III as 10 ml aliquots of taking a time of 4 minutes between each application.
  Arms: Experimental

SUMMARY:
This is a randomized controlled trial in which the safety and feasibility of cell therapy medicinal product shall be measured by comparing the variables of the response after treatment compared to baseline prior to implementation. Secondarily the results obtained are compared with each of the study groups.

Patients will receive concomitant basic pharmacological treatment for maintaining liver function.

All patients will be equally medically treated. The hypothetic test is to propose mononuclear cells from the bone marrow infused in the territory hepatic portal remaining segments (II and III) to be performed while contralateral portal embolization provides progenitor cells hepatic regenerative capacity that would shorten the time of liver regeneration and increase residual volume, facilitating the realization of an extended hepatectomy with greater assurance of maintaining proper residual function and adequate surgical margins.

DETAILED DESCRIPTION:
The study population corresponds to patients with hepatic space occupying lesion that require extended hepatic resection and in which the residual liver volume is insufficient to ensure liver function as well as required safety margins after resection.

The study population will consist of a total of 65 patients divided into two groups:

Study group: patients with hepatic space occupying lesion requiring an extended hepatic resection to those who are undergoing preoperative embolization segments portal intraportal affections and application of bone marrow cells.

Control group: patients with hepatic space occupying lesion that require an extended liver resection and who were performed preoperatively embolization portal of the affected segments.

The distribution of cases / controls will be 1/1. Patients in study group before surgery as well as portal embolization of the affected by the injury, will receive the experimental treatment being tested. Autologous bone marrow will be extracted by aspiration of the iliac crest under local anesthesia, and then the mononuclear cells (mo-MNCs) will be separated by density gradient centrifugation on Ficoll by an automatic procedure in the Laboratory for Cell Therapy.

In the control group patients will be held an embolization of liver segments in which are located the lesion.

It is estimated that the inclusion period is approximately 24 months plus the follow-up of each patient twelve months. Thus the total duration of the study will be about thirty-six months from the entry of the first patient until the end of the monitoring period of the last patient included.

The main objective is to evaluate the safety and feasibility of autologous bone marrow mononuclear cells as autologous liver regeneration enhancer, administered intraportal before surgery in patients with liver space occupying lesion that require extended hepatic resection and in which the residual liver volume is insufficient to ensure liver function and safety margins required after the resection.

Secondary objectives:

* Complications from regenerative therapy and / or study procedures.
* Increased volume obtained after applying the procedures of liver regeneration after surgery.
* The percentage of resections that has allowed liver regeneration.
* The liver functional status after surgery.
* The resection margins free of tumor.

Evaluation Methods:

Radiological assessment of liver volumes. Analytical evaluation of markers of regeneration.

ELIGIBILITY:
Inclusion Criteria:

1. - Patients of both sexes aged ≥ 18 years.
2. - Standard analytical parameters, defined by:

   * Leukocytes ≥ 3000
   * Neutrophils ≥ 1500
   * Platelets ≥ 100,000
   * Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) ≤ 1.5 standard range institution
   * creatinine ≤ 1.5 mg / dl
3. - Patients with liver space occupying lesion (LOE) that require extended hepatic resection.

Patient selection should be cautious, covering basically 5 types of liver damage which must be submitted prior to liver volumetry:

* Metastatic Disease subsidiary right hepatectomy extended to segment IV
* Metastatic Disease subsidiary right hepatectomy with suspected diseased liver (neoadjuvant chemotherapy) (in cases of doubt may be used liver function test "indocyanine green")
* Bilobar liver metastases with multiple nodules in the right lobe and more than 3 nodules greater than 30 mm in the left hepatic lobe (LHI) will perform lumpectomies the LHI + right portal branch ligation (or postoperative percutaneous embolization) in order to make right hepatectomy 4-6 weeks ("two stage" surgery)
* Subsidiary Hepatocarcinoma extended right hepatectomy
* Liver Injury benign / malignant (Hemangiomas, hydatid cysts or liver tumors / primary bile hepatoblastoma), which by extension threatens the viability of the remaining liver tissue.

  4 - Patients give their written informed consent for participation in the study and provide sufficient guarantees adherence to protocol according to the opinion of the investigator in charge of the patient care.

Exclusion Criteria:

1. Different tumor records current disease or any disease hematologic.
2. Patients with uncontrolled hypertension.
3. Severe heart failure (NYHA IV).
4. Patients with malignant ventricular arrhythmias or unstable angina.
5. Diagnosis of deep vein thrombosis in the previous 3 months.
6. Adjunctive therapy including hyperbaric oxygen, vasoactive substances, agents or angiogenesis inhibitors against Cox-II.
7. BMI> 40 kg/m2.
8. Patients with alcoholic with active alcoholism.
9. Proliferative retinopathy.
10. Concomitant disease that reduces life expectancy to less than a year.
11. Difficulty in monitoring.
12. Heart failure or ejection fraction (EF) <30%.
13. Stroke or myocardial infarction within the last 3 months.
14. Pregnant women or women of childbearing age who do not have adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-03; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events | 6 after drug administration of cell therapy.
  First 24 hours after administration of the mo-MNC, and monitoring at weeks 2,4 and 6 after drug administration of cell therapy.

SECONDARY OUTCOMES:
Changes in volume hepatic after application of hepatic regeneration procedures before surgery. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Padillo, MD, Principal Investigator — Head of General and Digestive Surgery, University Hospital Virgen del Rocio; Antonio Galindo, MD, Principal Investigator — Head of General and Digestive Surgery, University Hospital Nuestra Señora de Valme; Daniel Garrote, MD, Principal Investigator — Section Chief of General Surgery, University Hospital Virgen de las Nieves; Sebastian Rufian, MD, Principal Investigator — Head of General and Digestive Surgery, University Hospital Reina Sofia; Francisco Javier Padillo, MD, Study Chair — Head of General and Digestive Surgery, University Hospital Virgen del Rocio
Locations (1):
- University Hospital Virgen del Rocio, Seville, Sevilla, Spain

REFERENCES:
- See also: Andalusian Molecular Biology and Regenerative Medicine Centre — http://www.cabimer.es